CLINICAL TRIAL: NCT02857270
Title: A Phase 1 Study of an ERK1/2 Inhibitor (LY3214996) Administered Alone or in Combination With Other Agents in Advanced Cancer
Brief Title: A Study of LY3214996 Administered Alone or in Combination With Other Agents in Participants With Advanced/Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16419; I8S-MC-JUAB (Other: Eli Lilly and Company); 2016-001907-21 (EudraCT Number)
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Advanced Cancer; Metastatic Melanoma; Metastatic Non-small Cell Lung Cancer; Colorectal Cancer
Keywords: MAPK; RAS; BRAF
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — LY3214996; Midazolam; abemaciclib; 130-nm albumin-bound paclitaxel; Gemcitabine; encorafenib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- LY3214996 Dose Escalation (Experimental): LY3214996 given orally once a day (or twice a day) for 21 days.
  Interventions: Drug: LY3214996
- LY3214996 + Midazolam (Experimental): (Preliminary Drug-Drug Interactions [DDI])
  LY3214996 given orally (once a day) and midazolam given orally on cycle 1 day 1 and cycle 1 day 16 (21 day cycles except cycle 1 only = 22 days).
  Interventions: Drug: LY3214996; Drug: Midazolam
- LY3214996 Dose Expansion (Experimental): LY3214996 given orally (once a day) during each 21 day cycle.
  Interventions: Drug: LY3214996
- LY3214996 + Abemaciclib (Experimental): Dose Escalation and Expansion- LY3214996 given orally (dose timing will be determined) and abemaciclib given orally (single dose given during lead in period) twice a day every 12 hours during 21 day cycle.
  Interventions: Drug: LY3214996; Drug: Abemaciclib
- LY3214996 + Nab-Paclitaxel + Gemcitabine (Experimental): Dose Escalation and Expansion- LY3214996 given orally (dose timing will be determined) and nab-paclitaxel given intravenously (IV) on day 1, 8, and 15 and gemcitabine IV on day 1, 8, and 15 during each 28 day cycle.
  Interventions: Drug: LY3214996; Drug: Nab-paclitaxel; Drug: Gemcitabine
- LY3214996 + Encorafenib + Cetuximab (Experimental): Dose Escalation and Expansion- LY3214996 given orally, encorafenib given orally and cetuximab given IV.
  Interventions: Drug: LY3214996; Drug: Encorafenib; Drug: Cetuximab
- Japan Part 1 (Experimental): LY3214996 given orally.
  Interventions: Drug: LY3214996
- Japan Part 2 (Experimental): LY3214996 given orally and abemaciclib given orally.
  Interventions: Drug: LY3214996; Drug: Abemaciclib

INTERVENTIONS:
Drug: LY3214996 — Administered orally
Drug: Midazolam — Administered orally
  Arms: LY3214996 + Midazolam
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Japan Part 2; LY3214996 + Abemaciclib
Drug: Nab-paclitaxel — Administered IV
  Arms: LY3214996 + Nab-Paclitaxel + Gemcitabine
Drug: Gemcitabine — Administered IV
  Arms: LY3214996 + Nab-Paclitaxel + Gemcitabine
Drug: Encorafenib — Administered orally
  Arms: LY3214996 + Encorafenib + Cetuximab
Drug: Cetuximab — Administered IV
  Arms: LY3214996 + Encorafenib + Cetuximab

SUMMARY:
The purpose of this study is to determine the safety of an extracellular signal regulated kinase (ERK1/2) inhibitor LY3214996 administered alone or in combination with other agents in participants with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have advanced or metastatic cancer (solid tumors) and be an appropriate candidate for experimental therapy.

  * Part B (No Longer Enrolling Participants): Have advanced or metastatic cancer with an activating mitogen-activated protein kinase pathway alteration, BRAF mutant metastatic melanoma refractory to or relapsed after treatment with RAF and/or MEK inhibitors, metastatic melanoma with a NRAS mutation, or BRAF mutant NSCLC.
  * Part C: Advanced, unresectable cancer (dose escalation) and advanced, unresectable, or metastatic non-small cell lung cancer with a BRAF or RAS mutation, or NRAS mutant melanoma (dose expansion).
  * Part D (No Longer Enrolling Participants): Have metastatic pancreatic ductal adenocarcinoma (dose escalation and dose expansion).
  * Part E: Metastatic BRAF V600E colorectal cancer.
* Have discontinued previous treatments for cancer and have resolution, except where otherwise stated in the inclusion criteria, of all clinically significant toxic effects of prior chemotherapy, surgery, or radiotherapy to Grade ≤1 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0.
* Have adequate organ function.
* Have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) scale.

Exclusion Criteria:

* Have serious preexisting medical conditions.
* Have a known human immunodeficiency virus (HIV) infection or known activated/reactivated hepatitis A, B, or C.
* Have symptomatic central nervous system malignancy or metastasis.
* Have current hematologic malignancies, acute or chronic leukemia.
* Have a second primary malignancy that in the judgment of the investigator or Lilly may affect the interpretation of results.
* Have prior malignancies. Participants with carcinoma in situ of any origin and participants with prior malignancies who are in remission and whose likelihood of recurrence is very low, as judged by the Lilly clinical research physician, are eligible for this study.
* Have a mean QT interval corrected for heart rate (QTc) of ≥470 milliseconds on screening electrocardiogram (ECG) as calculated using the Bazett's formula at several consecutive days of assessment.
* Have participated, within the last 28 days in a clinical trial involving an investigational product or are currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have previously completed or withdrawn from this study or any other study investigating an ERK1/2 inhibitor.
* If female, is pregnant, breastfeeding, or planning to become pregnant.
* Have history or findings of central or branch retinal artery or venous occlusion with significant vision loss or other retinal diseases that cause current visual impairment or would likely cause visual impairment over the time period of the study.
* Currently using concomitant medications that are strong inhibitors or inducers of CYP3A4.
* Part C: have serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study, including interstitial lung disease (ILD) or severe dyspnea at rest or requiring oxygen therapy.
* Part C4 NRAS Melanoma: have previously completed or withdrawn from a study investigating a MEK inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with LY3214996 Dose Limiting Toxicities (DLTs) | Cycle 1 (21 Days)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration-Time Curve (AUC) of LY3214996 Administered as Monotherapy and when Administered in Combination with Nab-Paclitaxel Plus Gemcitabine, Abemaciclib and Encorafenib Plus Cetuximab | Cycle 1 Day 1 through Cycle 2 Day 1 (up to 28 Day Cycles)
PK: AUC of Gemcitabine when Administered with LY3214996 | Cycle 1 Day 1 through Cycle 1 Day 15 (28 Day Cycles)
PK: AUC of Nab-Paclitaxel when Administered with LY3214996 | Cycle 1 Day 1 through Cycle 1 Day 15 (28 Day Cycles)
PK: AUC of Abemaciclib and its Metabolites when Administered with LY3214996 | Cycle 1 Day 1 through Cycle 2 Day 1 (up to 22 Day Cycles)
PK: AUC of Encorafenib when Administered with LY3214996 | Cycle 1 Day 1 through Cycle 2 Day 1 (up to 22 Day Cycles)
PK: AUC of Cetuximab when Administered with LY3214996 | Cycle 1 Day 1 through Cycle 2 Day 1 (up to 22 Day Cycles)
PK: AUC of Midazolam and its 1'-Hydroxymidazolam Metabolite when Administered Alone and in Combination with LY3214996 | Cycle 1 Day 1 through Cycle 1 Day 16 (21 Day Cycles)
Objective Response Rate (ORR): Percentage of Participants With a Complete (CR) or Partial Response (PR) | Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Estimated up to 6 Months)
Duration of Response (DoR) | Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression or Death Due to Any Cause (Estimated up to 12 Months)
Time to First Response (TTR) | Baseline to Date of CR or PR (Estimated up to 6 Months)
Progression Free Survival (PFS) | Baseline to Progressive Disease or Death of Any Cause (Estimated up to 12 Months)
Disease Control Rate (DCR): Percentage of Participants who Exhibit Stable Disease (SD), CR or PR | Baseline through Measured Progressive Disease (Estimated up to 6 Months)
Overall Survival (OS) (Dose Expansion Arms Only) | Baseline to Date of Death from Any Cause (Estimated up to 2 Years)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (8):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - St Vincent's Hospital, Sydney, New South Wales
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- Gustave Roussy, Villejuif, France
- Japan (2):
  - Shizuoka Cancer Center, Sunto-Gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhagwat SV, McMillen WT, Cai S, Zhao B, Whitesell M, Shen W, Kindler L, Flack RS, Wu W, Anderson B, Zhai Y, Yuan XJ, Pogue M, Van Horn RD, Rao X, McCann D, Dropsey AJ, Manro J, Walgren J, Yuen E, Rodriguez MJ, Plowman GD, Tiu RV, Joseph S, Peng SB. ERK Inhibitor LY3214996 Targets ERK Pathway-Driven Cancers: A Therapeutic Approach Toward Precision Medicine. Mol Cancer Ther. 2020 Feb;19(2):325-336. doi: 10.1158/1535-7163.MCT-19-0183. Epub 2019 Nov 19. PMID 31744895
- See also: A Study of LY3214996 Administered Alone or in Combination With Other Agents in Participants With Advanced/Metastatic Cancer — https://trials.lillytrialguide.com/en-US/trial/64K6fy9q0Mw2eU8WyW2u4K